CLINICAL TRIAL: NCT01588275
Title: Cost-effectiveness of obstRuctivE Sleep Apnea Therapy (REST Study): Comparison of MRA Therapy Versus CPAP Therapy in Moderate OSAS
Brief Title: MRA Therapy Versus CPAP Therapy in Moderate OSAS
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: VitalAire Nederland BV (Unknown); SomnoMed Goedegebuure (Unknown)
Responsible Party: Principal Investigator, Grietje E de Vries, MSc, researcher/project leader, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL34138.042.10
Record Dates: First submitted 2012-04-25; First posted 2012-04-30 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Sleep Apnea, Obstructive
Keywords: cost-effectiveness; effectiveness; treatment; CPAP; MRA; compliance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance | interventions — Magnetic Resonance Angiography; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRA therapy (Active Comparator): During 12 months patients will be treated with a bibloc MRA (SomnoDent® MAS, SomnoMed Australia/Europe AG). The MRA will be customized by certified dentists or dental-specialists experienced in the field of dental sleep medicine.
  Interventions: Device: mandibular repositioning appliance (MRA) (SomnoDent)
- CPAP therapy (Active Comparator): During 12 months patients will be treated with Continuous positive airway pressure (CPAP).Treatment with CPAP prevents upper airway collapse by pneumatically "splinting" the upper airway during sleep.
  Interventions: Procedure: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: mandibular repositioning appliance (MRA) (SomnoDent) — bibloc MRA type SomnoDent starting at 70% protrusion of the mandibula
  Other Names: bibloc SomnoDent
  Arms: MRA therapy
Procedure: Continuous positive airway pressure (CPAP) — Proper CPAP-pressure will be set for each patient separately.
  Arms: CPAP therapy

SUMMARY:
The purpose of this study is to compare the cost-effectiveness and effectiveness of mandibular repositioning appliance (MRA) versus Continuous positive airway pressure (CPAP) therapy in patients with moderate Obstructive Sleep Apnea Syndrome (OSAS).

DETAILED DESCRIPTION:
Study design: In a randomized parallel controlled study 86 patients will be randomly assigned to either MRA therapy or CPAP therapy. Group A receives MRA. Group B receives CPAP. The total duration of the study is 12 months. Measurements will be done at baseline, after 3, 6 and 12 months.

Intervention: Group A will be treated with a bibloc MRA (Somnodent). The mandible will be set at 70% of the patient's maximum advancement and will be adjusted to the convenience of the patient. Titration will be continued until symptoms abate or until further advancement causes discomfort.

Group B will be treated with CPAP. Proper CPAP-pressure will be set for each patient separately. Patients are fitted with a comfortable CPAP mask before titration of the CPAP-pressure. For CPAP-titration, patients are instructed to adopt their own typical sleeping habits.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been subjected to polysomnography and are diagnosed as having moderate (AHI 15-30) OSAS;
* Aged ≥ 18 years;

Exclusion Criteria:

Medical and psychological criteria:

* Patients previously treated for OSAS (e.g. CPAP, MRA);
* Morphologic abnormalities of the upper airway (e.g., a compromised nasal passage, enlarged tonsils or adenoids, or upper airway soft-tissue or craniofacial abnormality);
* Reported or documented unstable endocrine dysfunction (hypothyroidism, acromegaly, or pituitary adenoma); Reported or documented severe cardiovascular- or pulmonary co-morbidity
* Clinically concurrent cardiovascular disease (coronary artery disease, heart failure,cardiac arrhythmias)
* CVA within 6 months prior to randomisation
* Daytime respiratory insufficiency
* Severe Chronic Obstructive Pulmonary Disease (COPD) (GOLD 3 or 4; FEV1 / FVC < 70% and FEV1 < 50%);
* Other diseases that may impact the evaluation of the results of the study according to the investigator's judgement.
* Reported or documented psychological condition precluding informed consent (e.g., mental retardation, depression or schizophrenia);

Whether the patient has unstable endocrine dysfunction, severe cardiovascular- or pulmonary co-morbidity or a psychological condition precluding informed consent, will be assessed by evaluating the patient's medical record.

Dental exclusion criteria:

* Extensive periodontal disease or tooth decay;
* Active temporomandibular joint disease (including severe bruxism);
* Restrictions in mouth opening (< 25mm) or advancement of the mandible <5mm);
* Partial or complete edentulism (less than eight teeth in upper or lower jaw).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-05-24 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Incremental cost-effectiveness ratio (ICER) in terms of AHI reduction and quality adjusted life years | 12 months
  Incremental cost-effectiveness ratio (ICER) in terms of AHI reduction measured during polysomnography and quality adjusted life years (QALYs)

SECONDARY OUTCOMES:
Change in quality of life | 3, 6 and 12 months
  EQ5D, SF-36, FOSQ questionnaires at baseline and after 3, 6 and 12 months
Change in Cardiovascular risk | 6 and 12 months
  smoking status, change from baseline ambulant blood pressure measurements after 12 months, blood samples, urine sample, accumulation of advanced glycation endproducts (AGEs) in skin tissue
Change in polysomnographic outcomes | 3 and 12 months
  total sleep time, sleep efficiency, minimal oxyhemoglobin saturation, arousals, sleep stages
Change in activities of daily living | 3 and 12 months
  Total distance on 6 minutes walking test Number of steps measured with pedometer
Compliance | 3, 6 and 12 months
  objective compliance by reading out devices subjective compliance by questionnaire
Side effects | 3, 6 and 12 months
  self-reported side effects from device dental and maxillofacial side-effects from both MRA and CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Grietje E de Vries, MSc, Study Chair — University Medical Center Groningen; Peter J Wijkstra, PhD, Principal Investigator — University Medical Center Groningen
Locations (3):
- Netherlands (3):
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - University Medical Center Groningen, Groningen
  - Martini Ziekenhuis Groningen, Groningen

REFERENCES:
- [Derived] Uniken Venema JAM, Knol-de Vries GE, van Goor H, Westra J, Hoekema A, Wijkstra PJ. Cardiovascular and metabolic effects of a mandibular advancement device and continuous positive airway pressure in moderate obstructive sleep apnea: a randomized controlled trial. J Clin Sleep Med. 2022 Jun 1;18(6):1547-1555. doi: 10.5664/jcsm.9908. PMID 35088708
- [Derived] de Vries GE, Hoekema A, Claessen JQPJ, Stellingsma C, Stegenga B, Kerstjens HAM, Wijkstra PJ. Long-Term Objective Adherence to Mandibular Advancement Device Therapy Versus Continuous Positive Airway Pressure in Patients With Moderate Obstructive Sleep Apnea. J Clin Sleep Med. 2019 Nov 15;15(11):1655-1663. doi: 10.5664/jcsm.8034. PMID 31739856
- [Derived] de Vries GE, Hoekema A, Vermeulen KM, Claessen JQPJ, Jacobs W, van der Maten J, van der Hoeven JH, Stegenga B, Kerstjens HAM, Wijkstra PJ. Clinical- and Cost-Effectiveness of a Mandibular Advancement Device Versus Continuous Positive Airway Pressure in Moderate Obstructive Sleep Apnea. J Clin Sleep Med. 2019 Oct 15;15(10):1477-1485. doi: 10.5664/jcsm.7980. PMID 31596213